CLINICAL TRIAL: NCT05485558
Title: Clinical Study Evaluating the Safety and Efficacy of N-acetyl Cysteine in Children With Drug-Resistant Epilepsy
Brief Title: the Safety and Efficacy of N-acetyl Cysteine in Children With Drug-Resistant Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amira Roshdy, Assistant Lecturer of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAC in DRE.
Record Dates: First submitted 2022-07-30; First posted 2022-08-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Drug Resistant Epilepsy
Keywords: N-acetyl cysteine
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): 30 patients will receive standard antiepileptic drug plus placebo capsules for 6 months.
  Interventions: Drug: Placebo
- N-acetyl cysteine group (Active Comparator): 30patients will receive 10 mg/kg of N-acetyl cysteine capsules together with their standard antiepileptic drug for 6 months.
  Interventions: Drug: N-acetyl cysteine
- N-actyl cysteine group (Active Comparator): 30 patients will receive 40 mg/kg of N-acetyl cysteine capsules together with their standard antiepileptic drug for 6 months.
  Interventions: Drug: NAc

INTERVENTIONS:
Drug: N-acetyl cysteine — 10 mg/kg of N-acetyl cysteine capsules together with their standard antiepileptic drug for 6 months.
  Other Names: NAC
  Arms: N-acetyl cysteine group
Drug: Placebo — 15 patients will receive standard antiepileptic drug plus placebo capsules for 6 months.
  Other Names: control
  Arms: Control group
Drug: NAc — 40 mg/kg of N-acetyl cysteine capsules together with their standard antiepileptic drug for 6 months.
  Arms: N-actyl cysteine group

SUMMARY:
This study aims at investigating the possible efficacy and safety of N-acetyl cysteine as adjuvant therapy in the treatment of drug-resistant epilepsy

DETAILED DESCRIPTION:
N-acetyl-cysteine (NAC), a glutathione precursor, is proven to activate the nuclear factor E2-related factor 2( Nrf2) in mouse models of status epilepticus, thus inhibiting high mobility group box 1 (HMGB1) cytoplasmic translocation in the hippocampal neural and glial cells and preventing the linkage between oxidative stress and neuroinflammation for which the redox-sensitive protein HMGB1 is central. Therefore,It may be useful as an adjuvant in treating various medical conditions, especially neuropsychiatry.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3-18 years with intractable childhood-onset epilepsy.

  * All patients are diagnosed to have drug-resistant epilepsy (refractory epilepsy) according to the ILAE definition.
  * The subject is willing and able to comply with the study requirements

Exclusion Criteria:

* Any metabolic conditions that might increase the risks associated with trial participation or investigational product administration, such as hepatic enzyme elevation greater than twice normal and/or a GFR < 60 mL/min/1.73 m2 or electrolyte imbalance.

  * Patients with Known allergy to N-acetyl cysteine.
  * Patients taking antioxidant and/or anti-inflammatory medications

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
effectivness of acetyl cysteine for controlling epileptic seizures in children with drug resistant epilepsy. | 6 months
  effectivness can be defined as more than 50% reduction in number of seizures.

SECONDARY OUTCOMES:
analyze the differences of improvement of quality of life via using Helth related quality of life questionnaire | 6 months
  Caregivers will complete the Quality of Life in Childhood Epilepsy (QOLCE) Scale(QOLCE-55).The QOLCE-55 sections' included the following domains: cognitive, emotional, social, and physical functioning Each item is on a 6-point Likert scale and includes anchors that are subjectively rated based on perceived QOL (e.g., 1 = very often, 2 = fairly often, 3 = sometimes, 4 = almost never, 5 = never, 6 = non-applicable).
  Caregivers completed the Quality of Life in Childhood Epilepsy (QOLCE) Scale.17

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed kishk, Lecturer, Study Director — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No